CLINICAL TRIAL: NCT02553278
Title: Clinical Study to Evaluate the Performances of Modified VelaShape and the Performance of Contour I V3 Devices for Abdominal Fat Reduction vs. Control
Brief Title: VelaShape and Contour I V3 for Abdominal Fat Reduction vs. Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHF18521
Record Dates: First submitted 2015-09-10; First posted 2015-09-17 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Unwanted Abdomen Fat
Keywords: abdominoplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment with VelaShape device (Experimental): One treatment will be performed by the VelaShape device on one randomized abdominal subarea, while the other abdominal subarea will not be treated and will serve as a control. Biopsies will be harvested during abdominoplasty and cultured. Two histology samples, for each subject, will be obtained during the abdominoplasty surgery, The arm is divided to 6 sub-groups, where each Sub-group contains up to 2 subjects as follows:
  Sub-group 1: Surgery immediately after treatment Sub-group 2: Surgery 5 days after treatment Sub-group 3: Surgery 10 days after treatment Sub-group 4: Surgery 20 days after treatment Sub-group 5: Surgery 30 days after treatment Sub-group 6: Surgery 60 days after treatment Sub-group 7: Surgery 90 days after treatment
  Interventions: Device: VelaShape device
- Treatment with Contour I V3 device (Experimental): One treatment will be performed by Contour I V3 device on one randomized abdominal subarea, while the other abdominal subarea will not be treated and will serve as a control. Biopsies from treated and untreated subareas will be harvested during abdominoplasty and cultured. Two histology samples, for each subject, will be obtained during the abdominoplasty surgery. The arm is divided to 6 sub-groups, where each Sub-group contains up to 2 subjects as follows:
  Sub-group 1: Surgery immediately after treatment Sub-group 2: Surgery 10 days after treatment Sub-group 3: Surgery 20 days after treatment Sub-group 4: Surgery 30 days after treatment Sub-group 5: Surgery 60 days after treatment Sub-group 6: Surgery 90 days after treatment
  Interventions: Device: Contour I V3 device

INTERVENTIONS:
Device: VelaShape device — Modified VelaShape radiofrequency device for non invasive fat reduction treatment.
  Arms: Treatment with VelaShape device
Device: Contour I V3 device — Contour I V3 device are non invasive for fat reduction.
  Arms: Treatment with Contour I V3 device

SUMMARY:
Prospective, 2-arm, clinical study for the evaluation of the VelaShape device and Contour I V3 device for non-invasive fat reduction vs. control.

All study subjects, who are scheduled for abdominoplasty, will undergo one treatment with VelaShape or Contour I V3 device.

Each arm will be treated with a different device:

Arm 1: subject will treated with VelaShape device Arm 2: subject will treated with Contour I V3 device

DETAILED DESCRIPTION:
Eligible subjects will undergo one treatment on one abdominal subarea. Another abdominal subarea will remain without treatment and will serve as a control. Biopsies from treated and untreated areas will be harvested during abdominoplasty and cultured.. Treatment with VelaShape will be performed to arm 1, and treatment with Contour I V3 will be performed to arm 2, according to the study protocol.

Each arm will be divided into 6 sub-groups, according to the following time interval between VelaShape or UltraShape treatment to surgery:

Sub-group 1: Surgery immediately after treatment Sub-group 2: Surgery 10 days after treatment Sub-group 3: Surgery 20 days after treatment Sub-group 4: Surgery 30 days after treatment Sub-group 5: Surgery 60 days after treatment Sub-group 6: Surgery 90 days after treatment Each Sub-group contains up to 2 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent to participate in the study.
2. Scheduled date for surgery (abdominoplasty).
3. Agree to provide samples for histology from the abdominoplasty.
4. Female and male subjects, between 18 to 60 years of age at the time of enrollment
5. Fitzpatrick Skin Type I to VI.
6. For Contour I V3 treatment only: Abdominal fat thickness of at least 1.5 cm (measured by calibrated caliper).
7. Female subjects must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
8. General good health confirmed by medical history and skin examination of the treated area.
9. Willing to follow the treatment and to provide histology samples during the surgery from the intended to be harvested areas.
10. Willingness to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
11. Willing to have photographs and images taken of the treated areas to be used (with de-identification) in evaluations, publications and presentations

Exclusion Criteria:

A subject is not eligible for participation in this study if he/she meets any of the following exclusion criteria:

1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, or abdominal aortic aneurism
2. Not intended to undergo surgery (abdominoplasty)
3. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
4. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
5. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
6. Having a permanent implant in the treated area, such as metal plates, or an injected chemical substance such as silicone
7. Having undergone any other surgery in the treatment area within 12 months of treatment or during the study, including liposuction
8. Previous body contouring procedures in the treatment area within 12 months
9. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing Known photosensitivity
10. Suffering from significant skin conditions in the treatment area or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course
11. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
12. Very poor skin quality (i.e., severe laxity)
13. Abdominal wall diastasis or hernia on physical examination
14. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
15. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
16. Unstable weight within the last 6 months (i.e., more than ± 3% weight change in the prior 6 months)
17. Participation in another clinical study within the last 6 months.
18. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-01-10 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
histology following VelaShape treatment | day 10 up to 90 days
  Evaluate abdominal fat reduction post VelaShape treatment vs.control
Histology following Contour I V3 treatment | day 10 up to 90 days
  Evaluate Abdominal fat reduction post Contour I V3 treatment vs. control

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Dean Ad-El, M.D, Principal Investigator — Plastic surgery department , Blinson - Rabin Hospital
Locations (1):
- Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Background] Adamo C, Mazzocchi M, Rossi A, Scuderi N. Ultrasonic liposculpturing: extrapolations from the analysis of in vivo sonicated adipose tissue. Plast Reconstr Surg. 1997 Jul;100(1):220-6. doi: 10.1097/00006534-199707000-00033. PMID 9207679